CLINICAL TRIAL: NCT03943017
Title: The Inspection Campaign of French Phase I/II Research Sites Following the BIA 10-2474 Accident: Medical vs. Regulatory Relevance
Brief Title: The Inspection Campaign of French Phase I/II Research Sites Following the BIA 10-2474 Accident
Acronym: HARMONY
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-08
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Health Knowledge, Attitudes, Practice; Safety Issues; Health, Subjective
Keywords: safety dysfunctions
MeSH Terms: conditions — Behavior | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Inspection and safety evaluation by 3 longstanding experience physicians of early clinical researches — Adjudicate each ARC's observations according to the 3 physicians perceived medical importance regarding safety; first, adjudications are performed separately. Then disagreements are settled during a final adjudication meeting between them.

SUMMARY:
Following the serious adverse events that occurred in January 2016 during the BIA 10 2474 First-in-Human study, the French Ministry of Health asked the Regional Health Agencies to inspect operations at all Authorized Research Centers (ARC) conducting phase I/II clinical trials of experimental drugs.

DETAILED DESCRIPTION:
Following the serious adverse events that occurred in January 2016 during the BIA 10 2474 First-in-Human study, the French Ministry of Health asked the Regional Health Agencies to inspect operations at all research sites conducting phase I/II clinical trials of experimental drugs.

All 30 sites of Île-de-France region fully authorized to perform phase I/II trials will be inspected by a physician and a public health pharmacist. Their reported list of observations will be submitted to three physicians with longstanding experience of early pharmacology studies performed in academic or private research facilities. These physicians will be asked to adjudicate each observation according to their perceived medical importance regarding safety. Adjudications will be first performed separately and disagreements will be later settled during a final adjudication meeting.

ELIGIBILITY:
Inclusion Criteria:

* Being one of the 30 sites of Île-de-France region fully authorized to perform phase I/II trials

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the 30 sites of Ile de France region fully authorized to perform phase I/II trials
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Number of observations which have potentially serious medical consequences after experts adjudication | Up to 2 years

SECONDARY OUTCOMES:
Number on disagreements occuring initially among the 3 adjudicators before adjudication | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Funck-Brentano, MD, PhD, Principal Investigator — INSERM, CIC-1421 and UMR ICAN 1166, Sorbonne Université, Faculty of Medicine, AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology and Clinical Investigation Center
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France